CLINICAL TRIAL: NCT00722813
Title: Cost Effectiveness and Utility of Coronary Artery Computed Tomography Angiography (CTA) in Screening for Coronary Artery Disease
Brief Title: Cost Effectiveness and Utility of Computed Tomography Angiography (CTA) and Cardiac Cath
Status: Completed | Type: Observational
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Aine Kelly, MD, Primary Investigator, University of Michigan
Other Study IDs: HUM00003409
Record Dates: First submitted 2008-07-24; First posted 2008-07-28 (Estimated); Last update posted 2013-11-21 (Estimated); Status verified 2013-11

CONDITIONS: Heart Diseases
MeSH Terms: conditions — Heart Diseases | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: Survey — To determine patient preference for the two tests CT angiography (CTA) and catheter coronary angiography (CCA).

SUMMARY:
This is a research study to determine patient preferences between two different diagnostic tests; a CT angiogram (CTA) and a catheter angiogram, both of which are used at the University to screen for and detect heart disease.

DETAILED DESCRIPTION:
This is a single site study that will retrospectively and prospectively identify and enroll 100 subjects, both male and female, 18 years of age and older who undergo both coronary angiography and coronary artery computed tomography (CT), using the electronic radiology and cardiology databases. The purpose is to conduct a survey to assess their preference for either test to diagnose coronary artery disease. Subjects should be within six months of having the tests to avoid memory and recall problems.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who have had both CTA and Coronary angiogram.
* 18 years old and older.

Exclusion Criteria:

* Under 18 years of age
* Memory Impairment:

  * Stroke
  * Traumatic brain Injury
  * Dementia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects who have had both CTA and Cardiac catherizations
Sampling Method: Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2006-10; Primary Completion 2012-10 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Utility of CT and catheter angiography | Within 6 months of testing with CT and catheter angiography
  Utility of CT and catheter angiography was compared within patients who had both tests performed.

CONTACTS AND LOCATIONS:
Overall Officials: Aine Kelly, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan Health Systems, Ann Arbor, Michigan, United States